CLINICAL TRIAL: NCT01385306
Title: Noninvasive Neurostimulation of the Vagus Nerve With the AlphaCore System for the Relief of Acute Bronchoconstriction Due to Asthma
Brief Title: Noninvasive Neurostimulation of the Vagus Nerve for the Relief of Acute Bronchoconstriction Due to Asthma
Acronym: BC-SA-01
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: ElectroCore INC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BC-SA-01
Record Dates: First submitted 2011-06-17; First posted 2011-06-30 (Estimated); Results first posted 2018-10-10 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AlphaCore System (Experimental): non-invasive vagus nerve stimulation (nVNS) using the AlphaCore System
  Interventions: Device: AlphaCore System

INTERVENTIONS:
Device: AlphaCore System — Non-invasive neurostimulation of the vagus nerve

SUMMARY:
The objective of this feasibility research study is to gather preliminary clinical data regarding the safety and potential clinical benefit of noninvasive neurostimulation of the vagus nerve with the AlphaCore™ system for the relief of acute bronchoconstriction due to asthma.

DETAILED DESCRIPTION:
The purpose of the study was to collect initial safety and efficacy information of use of the AlphaCore System by clinicians in an emergency setting as an adjunctive treatment to standard of care for the relief of acute bronchoconstriction. After consent was obtained and screening completed, subjects were stimulated two times, 30 minutes apart, for 90 seconds each. Subjects were assessed prior to and immediately post the first stimulation and at 15, 30, 60, and 90 minutes; follow was also conducted at day 7 and day 30.

ELIGIBILITY:
Inclusion Criteria:

1. Is between the ages of 18 and 70 years.
2. Has been admitted to an emergency care facility with a working diagnosis of bronchoconstriction due to asthma.
3. Has an FEV1<60% predicted.
4. Is available and willing to return for an office visit at 7 days and participate in a 30-day telephone call from time of discharge from the ED.
5. Is able to give written Informed Consent, or his/her legally authorized representative is available to give written Informed Consent.

Exclusion Criteria:

1. Has a history of lung cancer, chronic obstructive pulmonary disease (COPD), or other co-morbidity due to irreversible narrowing of the airways.
2. Is at risk of imminent respiratory collapse:

   * Lung Function: FEV1 < 25% predicted
   * Signs and symptoms of extreme respiratory distress at rest, such as accessory muscle use, chest retraction
   * Consciousness State: Drowsy, confused
   * Rapid deterioration in respiratory status (sudden change in respiratory rate, decrease in oxygen saturation, change in consciousness, etc).
3. Has an abscess or other infection or lesion (including lymphadenopathy) at the therapy head placement site.
4. Has known or suspected atherosclerotic cardiovascular disease, carotid artery disease (e.g. bruits or history of TIA or CVA) or congestive heart failure (CHF).
5. Has suspected or confirmed sepsis.
6. Has a clinically significant irregular heart rate or rhythm.
7. Clinically significant changes in blood pressure or is receiving pressors to maintain blood pressure.
8. Is currently implanted with an electrical and/or neurostimulator device, including but not limited to cardiac pacemaker, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator, or cochlear implant.
9. Has a history of carotid endarterectomy or vascular neck surgery on the right side.
10. Has been implanted with metal cervical spine hardware.
11. Has a condition that would interfere with VAS Dyspnea self-assessment.
12. Is pregnant.
13. Is participating in any other therapeutic clinical investigation or has participated in a clinical trial in the preceding 30 days.
14. Belongs to a vulnerable population or has any condition such that his or her ability to provide informed consent, comply with follow-up requirements, or provide self-assessments is compromised (e.g., homeless, developmentally disabled, prisoner).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elmin Steyn, MD, Principal Investigator; Zunaid Mohammed, MD, Principal Investigator — unafiliated; Robert Johnson, Principal Investigator — unafiliated; Dale Cilliers, Principal Investigator — unafiliated
Locations (5):
- South Africa (5):
  - Kuilsriver Hospital, Kuils River, Cape Town
  - Panorama Mediclinic, Panorama, Cape Town
  - Life Vincent Pallotti Hospital, Pinelands, Cape Town
  - Cape Gate Medi-Clinic Hospital, Stellenbosch, Cape Town
  - Christiaan Barnard Memorial Hospital, Cape Town

REFERENCES:
- [Derived] Steyn E, Mohamed Z, Husselman C. Non-invasive vagus nerve stimulation for the treatment of acute asthma exacerbations-results from an initial case series. Int J Emerg Med. 2013 Mar 19;6(1):7. doi: 10.1186/1865-1380-6-7. PMID 23510361

RESULTS

PARTICIPANT FLOW:
Groups:
- AlphaCore System: Non-invasive Neurostimulation: AlphaCore System: Non-invasive neurostimulation of the vagus nerve
Period: Overall Study
Arm/Group | AlphaCore System: Non-invasive Neurostimulation
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Population
Arm/Group | AlphaCore System: Non-invasive Neurostimulation
Number analyzed (Participants) | 6
Age, Continuous [Mean (Full Range); unit: years] | 41 [32 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5
  Asian | 1
Region of Enrollment [Number; unit: participants]
  South Africa | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Subjects were assessed for adverse events for the duration of procedure. Subjects were also seen at 7 days and had a phone call at 30 days from the date of the stimulation procedure.
Time Frame: 30 days
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | AlphaCore System: Non-invasive Neurostimulation
Number analyzed (Participants) | 6
Participants | 2

2. Secondary Outcome: Number of Participants With a Change in FEV1 (Forced Expiratory Volume at 1 Second) of 12% or More From Baseline to 30 Minutes
Description: Improvement in FEV1 was defined as an increase of at least 12% compared with baseline (pre-first stimulation). The 30 minute measure was taken immediately after the second stimulation.
  (FEV1 measured as a percentage of normal, where greater that 80% is normal and less than 40% is severe degree of obstruction.)
Time Frame: 30 minutes
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | AlphaCore System: Non-invasive Neurostimulation
Number analyzed (Participants) | 6
Participants | 4

3. Secondary Outcome: Improvement in Dyspnea Score of at Least 1.5 Points From Baseline to 30 Minutes
Description: Improvement in dyspnea was defined as at least 1.5 point decrease on a 10 point Visual Analogue Scale (VAS) compared with baseline (pre-first stimulation). Where 0 = no dyspnea and 10 = very severe dyspnea. The 30 minute measure was taken immediately after the second stimulation.
Time Frame: 30 minutes
Population: Safety population
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | AlphaCore System: Non-invasive Neurostimulation
Number analyzed (Participants) | 6
units on a scale
  Dyspnea score Pre-stimulation | 6.75 [5.2 to 9.2]
  Dyspnea score at 30 minutes | 3.10 [0 to 4.4]

4. Secondary Outcome: Time to Discharge From the Emergency Department
Description: Time to discharge from the emergency department post stimulation
Time Frame: Duration of stay in emergency room - up to approximately 6 hours.
Population: Safety population.
Measure: Mean (Full Range); unit: minutes
Arm/Group | AlphaCore System: Non-invasive Neurostimulation
Number analyzed (Participants) | 6
minutes | 193 [100 to 294]

5. Secondary Outcome: Number of Participants With Requirement for Concomitant Medications
Description: Requirement for concomitant medications. Medications administered in the emergency department pre and post stimulation
Time Frame: Duration of stay in emergency room, up to approximately 6 hours
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | AlphaCore System: Non-invasive Neurostimulation
Number analyzed (Participants) | 6
Participants
  Pre stimulation medications | 5
  Post simulation medications | 6

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | AlphaCore System: Non-invasive Neurostimulation
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AlphaCore System: Non-invasive Neurostimulation (N=6)
Hospitalization for respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AlphaCore System: Non-invasive Neurostimulation (N=6)
Chest tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less